CLINICAL TRIAL: NCT06355934
Title: OverTTuRe: An Observational Multi-Country Study Collecting Real-World Secondary Data on the Characteristics, Treatment Patterns and Outcomes of Patients With ATTR Amyloidosis
Brief Title: OverTTuRe: Characteristics, Treatment Patterns and Outcomes of Patients With ATTR Amyloidosis
Acronym: OverTTuRe
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8450R00004
Record Dates: First submitted 2024-02-12; First posted 2024-04-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: ATTR Amyloidosis
Keywords: ATTR-CM, ATTRv-PN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (6):
- ATTR cardiomyopathy: Patients with Transthyretin Amyloidosis Cardiomyopathy
  Interventions: Other: no intervention
- ATTR polyneuropathy: Patients with Transthyretin Amyloidosis Neuropathy
  Interventions: Other: no intervention
- ATTR unknown: Patients with ATTR unknown genotype
  Interventions: Other: no intervention
- ATTR with mixed phenotype: Patients with ATTR mixed phenotype
  Interventions: Other: no intervention
- ATTR wild type: Patients with Transthyretin Amyloidosis wild type
  Interventions: Other: no intervention
- ATTR hereditary: Patients with Transthyretin Hereditary
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — not applicable, this is an observational retrospective data analysis study; no interventions in the study

SUMMARY:
The overall aim of this observational study is to generate real-world evidence on the pre- and post-diagnosis disease journeys, including baseline characteristics, treatment patterns and selected clinical, economic, and humanistic outcomes (for example Health Related Quality of Life (HRQoL), Neuropathy impairment score, activities of daily living (ADL) assessments) in patients with ATTR amyloidosis, and to better understand how the disease is presented.

DETAILED DESCRIPTION:
This retrospective, observational, longitudinal, multi-country cohort study aims to describe characteristics, treatment patterns, and outcomes in ATTR amyloidosis patients.

Primary objectives: Describe patient characteristics (for example demographics, family history of ATTR, key comorbidities and humanistic outcomes (e.g. Health Related Quality of Life (HRQoL), Neuropathy impairment score, activities of daily living (ADL) assessments), treatment patterns, and disease outcomes. Characterize and quantify the healthcare resource utilization (HCRU) in ATTR amyloidosis patients who will be followed post-index until the end of follow-up.

Secondary objectives: Describe demographics, clinical characteristics and HCRU in ATTR amyloidosis patients prior to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years at study index date AND
* A reported diagnosis code for amyloidosis OR
* A claim for ATTR-specific treatment OR
* A positive biopsy for amyloidosis and positive immunostaining result of biopsy for ATTR

Exclusion Criteria:

* Evidence of primary (AL) and secondary (AA) amyloidosis AND/OR
* At least one claim/procedure code for stem cell transplant or at least two claims/procedure codes for chemotherapy and autoimmune disease drugs which may represent AL (primary) or AA (secondary) amyloidosis treatments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include data from patients aged > 18 years with a diagnosis of ATTR amyloidosis or other evidence confirming ATTR amyloidosis. Patients will be followed until exit from the database (loss to follow-up), death, or end of database period (data collection). Baseline data will apply a lookback period of 12 months. Patient identification will be from 2014-01-01 onwards
Sampling Method: Non-Probability Sample
Enrollment: 55000 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Health Care Resource Utilization (HCRU) - Outpatient visits | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Annualized events rate for: Overall outpatient visits
Health Care Resource Utilization (HCRU) - Outpatient visits by specialty | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Annualized events rate for: Overall outpatient visits by specialty
Health Care Resource Utilization (HCRU) - Emergency department visits | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Annualized events rate for: Emergency department visits
Health Care Resource Utilization (HCRU) - Hospitalizations, length of stay | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Annualized events rate for: Hospitalizations (bed days)
Health Care Resource Utilization (HCRU) - Hospitalizations | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Annualized events rate for: Hospitalizations Overlaps (e.g., hospitalization after emergency department visit) are allowed and counted as separate visits
Health Care Resource Utilization (HCRU) - Health care cost | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  This variable will describe all-cause direct medical and pharmacy costs only, utilizing the amount charged, where available in the data. The direct medical costs will include costs incurred from inpatient stays, outpatient visits, emergency room visits, procedures, and laboratory tests. The inclusion of pharmacy costs is subject to data availability and will include all pharmacy costs per patient separated on pharmacy dispensed and in-hospital dispensed when possible. When feasible, costs will be divided on all-cause, CV, and other specialties
Cardiac transplant | From diagnosis of ATTR amyloidosis (index date) until date of first cardiac transplant, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Cardiac transplant (Time to event)
All cause mortality | From diagnosis of ATTR amyloidosis (index date) until date of death due to any cause, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Mortality (time-to-event)
Liver transplant | From diagnosis of ATTR amyloidosis (index date) until date of first liver transplant, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Liver transplant (time-to-event)
Heart Failure Hospitalization | From diagnosis of ATTR amyloidosis (index date) until date of first hospitalization for heart failure, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Heart failure hospitalization (time-to-event)
New ATTR amyloidosis clinical manifestation | From diagnosis of ATTR amyloidosis (index date) until date of first diagnosis of new ATTR amyloidosis clinical manifestation, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  New amyloidosis manifestation (time-to-event); Time to the first development of a new clinical manifestation that the patient did not have pre-index)
Hospitalization (any cause) | From diagnosis of ATTR amyloidosis (index date) until date of first hospitalization for any reason, assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Time to hospitalization (all-cause)
Neuropathy Impairment Score (NIS) | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  The NIS Score has a range of 0 to 244 and a higher NIS score indicates poorer function
Neuropathy Impairment Score Lower Limbs (NIS-LL) | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  The NIS-LL score has a range of 0-88 and a greater NIS-LL score indicates poorer function
Neuropathy Impairment Score +7 (NIS+7) | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  The NIS+7 Score has a range of -26.04 to 270.04 and a higher NIS+7 score indicates poorer function
Neuropathy Impairment Score modified +7 (mNIS+7) | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  The mNIS+7 Score has a range of -22.32 to 102.32 and a higher mNIS+7 score indicates poorer function
Neuropathy symptoms and change (NCS) score | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  NSC score is a questionnaire composed of 38 questions that assess the presence and severity of these neuropathy symptoms. The NSC score ranges from -114 to 114 for males and -108 to 108 for females. Greater scores indicate worse symptom severity; a negative value indicates an improvement in symptom severity from baseline
PND (Polyneuropathy Disability) | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  The PND is a 6-stage scoring system: Stage 0: no impairment; Stage 1: sensory disturbances but preserved walking capabilities; Stage 2: impaired walking capacity, but ability to walk without a stick or crutches; Stage 3A/B: walking with help of 1 or 2 sticks or crutches; Stage 4: confined to wheel chair or bedridden. A greater stage indicates greater impairment
Other relevant clinical measurement of ATTR amyloidosis functional status | From diagnosis of ATTR amyloidosis (index date), assessed throughout the study until end of follow-up, up to a maximum of 12 years
  Any other relevant clinical measurement of ATTR amyloidosis functional status

SECONDARY OUTCOMES:
Health Care Resource Utilization (HCRU) - Outpatient visits | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  Annualized events rate for: Overall outpatient visits
Health Care Resource Utilization (HCRU) - Outpatient visits by specialty | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  Annualized events rate for: Overall outpatient visits by specialty
Health Care Resource Utilization (HCRU) - Emergency department visits | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  Annualized events rate for: Emergency department visits
Health Care Resource Utilization (HCRU) - Hospitalizations, length of stay | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  Annualized events rate for: Hospitalizations (bed days)
Health Care Resource Utilization (HCRU) - Hospitalizations | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  Annualized events rate for: Hospitalizations Overlaps (e.g., hospitalization after emergency department visit) are allowed and counted as separate visits
Health Care Resource Utilization (HCRU) - Health care cost | From up to 12 years prior to ATTR amyloidosis diagnosis, assessed throughout the study, up to a maximum of 12 years.
  This variable will describe all-cause direct medical and pharmacy costs only, utilizing the amount charged, where available in the data. The direct medical costs will include costs incurred from inpatient stays, outpatient visits, emergency room visits, procedures, and laboratory tests. The inclusion of pharmacy costs is subject to data availability and will include all pharmacy costs per patient separated on pharmacy dispensed and in-hospital dispensed when possible. When feasible, costs will be divided on all-cause, CV, and other specialties

CONTACTS AND LOCATIONS:
Locations (26):
- Research Site, Eden Prairie, Minnesota, United States
- Research Site, Calgary, Alberta, Canada
- China (5):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Wuhan
- Research Site, Horsens, Denmark
- Research Site, Berlin, Germany
- Research Site, Tokyo, Japan
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Spain (11):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, El Palmar
  - Research Site, Huelva
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Palma de Mallorca
  - Research Site, Salamanca
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Södertälje
  - Research Site, Umeå
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Gillmore JD, Hahn K, Smith JG, Conceicao I, Tian Z, Grogan M, Pao C, Wittbrodt E, Jarbrink K, Papas MA, Davis MK. Rationale and Design of ANTHOLOGY: An ATTR Amyloidosis Real-World Evidence Program Aiming to Address Gaps in Amyloidosis Care. Cardiol Ther. 2025 Sep;14(3):477-490. doi: 10.1007/s40119-025-00402-y. Epub 2025 Mar 19. PMID 40108078